CLINICAL TRIAL: NCT06360484
Title: Prevalence and Clinical Characterization of Hepatitis D Virus (HDV) Infection Among Sudanese Patients With Hepatitis B Virus (HBV), A Cross-Sectional Study
Brief Title: Prevalence and Clinical Characterization of Hepatitis D Virus (HDV) Infection Among Sudanese Patients With Hepatitis B Virus
Status: Completed | Type: Observational
Sponsor: National Center for Gastroentestinal and Liver Disease (Other)
Responsible Party: Sponsor
Other Study IDs: PrevelanceHDVSudan
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Hepatitis B; Hepatitis D; Viral Hepatitis
MeSH Terms: conditions — Hepatitis B; Hepatitis D | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: investigations for Hepatitis D virus — Investigations included liver function tests, abdominal ultrasounds to identify features of chronic liver disease, and evidence of decompensation. ELISA for Ant-HDV-IgG was conducted.

SUMMARY:
Background: Sudan has a high prevalence of hepatitis B surface antigen (HBsAg), exceeding 8%. The prevalence of hepatitis B varies across different regions of Sudan, ranging from 6.8% in central Sudan to as high as 26% in southern Sudan. Hepatitis B virus (HBV) infection can lead to various complications, including cirrhosis, liver failure, and hepatocellular carcinoma (HCC). Hepatitis D virus (HDV) relies on HBV for replication and can accelerate the progression of HBV-related liver diseases, leading to more severe outcomes. This study aims to determine the prevalence of HDV infection among Sudanese patients with HBV-related liver diseases and to investigate the clinical characteristics of patients with HBV/HDV co-infection.

Design/Method: This descriptive cross-sectional hospital-based study was conducted at Ibn Sina Specialized Hospital in Sudan between June and September 2022. Ninety HBV patients aged 16 years and above were included. Patients were interviewed using a structured questionnaire, and medical histories and examinations were recorded. Investigations included liver function tests, abdominal ultrasounds, and ELISA for Ant-HDV-IgG

ELIGIBILITY:
Inclusion Criteria:

* patients aged 16 years and above
* with hepatitis B virus infection

Exclusion Criteria:

* patients with HIV or HCV co-infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was conducted between June and September 2022, involving patients aged 16 years and above with hepatitis B virus infection. Patients attending the liver clinic or admitted at Ibn Sina Specialized Hospital were included, while those with HIV and HCV co-infection were excluded.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
the prevalence of hepatitis D infection among Sudanese patients with HBV-related liver diseases. | June 2022 - September 2022
  to ascertain the prevalence of hepatitis D infection among Sudanese patients with HBV-related liver diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Gastrointestinal and Liver Diseases, Khartoum, Sudan